CLINICAL TRIAL: NCT06589427
Title: Prediction of PaO2 from SpO2 Values in Critically Ill Invasively Ventilated Patients - Rationale and Protocol for a Patient-level Analysis of ERICC, LUNG SAFE, PRoVENT and PRoVENT-iMiC (PRoPERLy II)
Brief Title: Prediction of PaO2 Values Using the PRoPERLy II Database
Acronym: PRoPERLy-II
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: PRoPERLy-II
Record Dates: First submitted 2024-07-22; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Invasive Ventilation
Keywords: Intensive care; Invasive ventilation; PaO2 prediction; Risk stratification; P/F; S/F
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Invasively ventilated intensive care unit patients.: Critically ill patients receiving invasive ventilation for various reasons, like ARDS, or AHRF.
  Interventions: Other: Invasive ventilation.

INTERVENTIONS:
Other: Invasive ventilation. — Patients were subjected to invasive ventilation.
  Other Names: Respiratory support.

SUMMARY:
Four prospective observational studies of ventilation in critically ill patients were harmonized and pooled.

DETAILED DESCRIPTION:
The individual data from four observational studies ('Epidemiology of Respiratory Insufficiency in Critical Care study' [ERICC], the 'Large Observational Study to Understand the Global Impact of Severe Acute Respiratory Failure' [LUNG SAFE], 'PRactice of VENTilation in critically ill patients without ARDS' [PRoVENT], 'PRactice of VENTilation in critically ill patients in Middle-income Countries' [PRoVENT-iMiC]) were harmonized and pooled into a database named 'PRoPERLy II'. This database will be used to address various issues in diverse patient categories.

ELIGIBILITY:
ERICC included patients aged 18 years or older that received ventilatory support for at least 24 hours during the first 48 hours of ICU admission at the participating ICUs. ERICC excluded patients with a tracheostomy, patients admitted for routine uncomplicated postoperative care, readmissions and patients with a terminal condition. ERICC enrolled patients during 2-months period.

LUNG SAFE included patients aged 16 years or older that received invasive or noninvasive ventilation. LUNG SAFE excluded patients without informed consent. LUNG SAFE enrolled patients during a 4-week period in the winter months.

PRoVENT included patients aged 18 years or older that received invasive ventilation. PRoVENT excluded patients in whom ventilation was started before the study recruitment week, patients receiving only noninvasive ventilation, and patients that were transferred to the ICU from another hospital under ventilation. PRoVENT enrolled patients during 4-week period.

PRoVENT-iMiC included patients aged 18 years or older that started with invasive ventilation. They excluded patients that received only noninvasive ventilation, patients whose invasive ventilation started before the inclusion phase of the study, and patients transferred from another hospital while under ventilation. PRoVENT-iMiC enrolled patients during 4-week period.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in the PRoPERLy II database are eligible for this and future analyses. For this first analysus, patients without reported SpO2 values and patients with SpO2 values and PaO2 values not simultaneously recorded are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Mortality. | ICU visit, anticipated average 4 days
  Mortality risk based on PaO2/FiO2 or SpO2/FiO2.

SECONDARY OUTCOMES:
Predicted PaO2. SpO 2 /FiO 2 ratios and of predicted PaO 2 /FiO 2 ratios. | In the first 4 days of invasive ventilation.
  PaO2 values predicted from SpO2 values.
Predicted PaO2/FiO2 SpO 2 /FiO 2 ratios and of predicted PaO 2 /FiO 2 ratios. | In the first 4 days of invasive ventilation.
  PaO2/FiO2 predicted from SpO2/FiO2

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, Principal Investigator — Amsterdam UMC
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
For this, interested investigators will have to provide a detailed analysis plan, containing a testable hypothesis, clearly described endpoints and an analysis plan. After approval, investigators will be provided with a mock database that will allow them to write an analysis script in R. PROVE network investigators will then run the script on the PRoPERLy II database and provide the investigators with the results. Any publication from an additional analysis must follow the rules for publication denoted by the PROVE network
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Notably, after this initial analysis of PRoPERLy II, the database will be available for additional analysis, till for ever
Access Criteria: For this, interested investigators will have to provide a detailed analysis plan, containing a testable hypothesis, clearly described endpoints and an analysis plan. After approval, investigators will be provided with a mock database that will allow them to write an analysis script in R. PROVE network investigators will then run the script on the PRoPERLy II database and provide the investigators with the results. Any publication from an additional analysis must follow the rules for publication denoted by the PROVE network
URL: https://www.provenetwork.org/